CLINICAL TRIAL: NCT01952262
Title: Ultrasound Evaluation of Diaphragmatic Dysfunction in Critically Ill Patients. An Observational Study.
Brief Title: Ultrasound of the Diaphragm in ICU Patients
Status: Completed | Type: Observational
Sponsor: Università Vita-Salute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Landoni, Head of Research, Università Vita-Salute San Raffaele
Other Study IDs: OSR/39/05/13
Record Dates: First submitted 2013-08-02; First posted 2013-09-27 (Estimated); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Critically Ill
Keywords: ultrasound; diaphragm; intensive care; critical care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- critically ill ICU patients: critically ill intensive care unit patients
  Interventions: Other: diaphragm ultrasound

INTERVENTIONS:
Other: diaphragm ultrasound — we'll perform diaphragm ultrasound in ICU critically ill patients
  Other Names: echography of diaphragm

SUMMARY:
Diaphragmatic dysfunction is an important complication of mechanical ventilation. Critically ill patients admitted in a teaching hospital intensive care unit will be evaluated with diaphragm ultrasound to investigate predictors of diaphragmatic dysfunction and the clinical course of these patients.

Vascular surgery patients (aortic abdominal surgery) might also be included and assessed with diaphragm ultrasound before and after surgery irrespectively of the need of intensive care unit. On December 2014 the Etical committee approved an amendment to include the possibility to study elective aortic abdominal surgery patient to assess the relationship between surgery related diaphragmatic dysfunction and postoperative respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* adult plus admitted in ICU plus invasive or non-invasive mechanical ventilation or
* adults aortic vascular surgery

Exclusion Criteria:

* < 18 years

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Diaphragmatic dysfunction | participants will be followed for the duration of intensive care unit stay, an expected average of 1 weeks
  Diaphragmatic dysfunction will be measured as thickness and inspiratory excursion of the diaphragm

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Zambon, MD, Principal Investigator — San Raffaele Scientific Institute
Locations (1):
- Ospedale San Raffaele di Milano, Milan, Italy